CLINICAL TRIAL: NCT03230799
Title: Comparison of Minimal Invasive Lens Surgery and Traditional Cataract Surgery for Treating Congenital Cataracts
Brief Title: Comparison of Minimal Invasive Lens Surgery and Traditional Cataract Surgery
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Sun Yat-sen University (Other)
Responsible Party: Principal Investigator, Haotian Lin, Clinical Professor, Sun Yat-sen University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: CCPMOH2017-China-3
Record Dates: First submitted 2017-07-17; First posted 2017-07-26 (Actual); Last update posted 2022-05-17 (Actual); Status verified 2022-04

CONDITIONS: Congenital Cataract
Keywords: congenital cataract; minimal invasive surgery; secondary intraocular lens implantation

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- traditional cataract surgery (Active Comparator): Central anterior continuous capsulorhexis (5-6 mm)+ irrigation/aspiration + posterior capsulorhexis + anterior vitrectomy（ACCC+ I/A + PCCC + Anti-vit)
  Interventions: Procedure: traditional cataract surgery
- minimal invasive lens surgery (Experimental): Peripheral capsulorhexis opening (1.0-1.5 mm)+irrigation/aspiration
  Interventions: Procedure: minimal invasive lens surgery

INTERVENTIONS:
Procedure: minimal invasive lens surgery — We decreased the size of the capsulorhexis opening to 1.0-1.5 mm in diameter. Then we moved the location of the capsulorhexis to the peripheral area of the lens instead of the central area. A 0.9 mm phacoemulsification probe was used to remove the lens contents and/or cortical opacities.
  Arms: minimal invasive lens surgery
Procedure: traditional cataract surgery — ACCC+ I/A + PCCC + Anti-vit: anterior continuous capsulorhexis + irrigation/aspiration + posterior capsulorhexis + anterior vitrectomy
  Arms: traditional cataract surgery

SUMMARY:
Previously, we have developed a minimal invasive lens surgery in the purpose of reduce post-operative complications of congenital cataract. This prospective, randomized controlled study aims at comparing the prognosis of the minimal invasive lens surgery and the traditional cataract surgery for treating congenital cataracts.

DETAILED DESCRIPTION:
Patients with congenital cataract that requires surgical intervention are enrolled. Then the patients are assigned to two groups: Group I: the participants receive a minimal invasive lens surgery, while in Group II, the participants receive a traditional cataract surgery. A secondary intraocular lens implantation is performed when the patient is two years old for both Group I and Group II. Investigators then compare the visual acuity, incidence of high intraocular pressure, incidence of visual axis opacification, uveitis and iris/pupil abnormality between two groups, to evaluate and compare the prognosis of minimal invasive lens surgery and traditional cataract surgery for treating congenital cataracts.

ELIGIBILITY:
Inclusion Criteria:

* Age between 1 month and 24 months
* Uncomplicated congenital cataract (≥ 3 mm central dense opacity) in one or both eyes with an intact non-fibrotic capsular bag
* Informed consent signed by a parent or legal guardian

Exclusion Criteria:

* confirmed or suspected hereditary cataract, including and not restricted to family history of congenital cataract
* Intraocular pressure >21 mmHg
* Preterm birth (<28 weeks)
* Presence of other ocular diseases (keratitis, keratoleukoma, aniridia, glaucoma) or systemic disease (congenital heart disease, ischemic encephalopathy)
* History of ocular diseases (any congenital eye diseases, such as, congenital cataract, congenital glaucoma, congenital aniridia) in the family
* History of ocular trauma
* Microcornea
* Persistent hyperplastic primary vitreous
* Rubella
* Lowe syndrome

Ages: 1 Month to 24 Months | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 100 (Estimated)
Dates: Start 2017-07-28 (Actual); Primary Completion 2022-06 (Estimated); Study Completion 2022-12 (Estimated)

PRIMARY OUTCOMES:
Best correctied visual acuity | recorded at each follow-up to five years of age.
  Determined with the Teller's acuity card, the Lea symbol visual acuity chart or the ETDRS chart according the patient's age.

SECONDARY OUTCOMES:
High intra-ocular pressure | after lens removal to five years of age.
  Determined with Tono-Pen tonometer at each follow-up
Visual axis opacification | after lens removal to five years of age.
  Determined with slit-lamp photography at each follow-up
Bi-ocular visual function | performed when the patient is four years old and five years old.
  Determined with synoptophore

CONTACTS AND LOCATIONS:
Overall Officials: Yizhi Liu, M.D,Ph.D, Principal Investigator — Zhongshan Ophthalmic Center, Sun Yat-sen University
Locations (1):
- Zhongshan Ophthalmic Center,Sun Yat-sen U, Guangzhou, Guangdong, China

IPD SHARING:
Plan to Share IPD: No